CLINICAL TRIAL: NCT03316833
Title: The ROLEX Registry (Revascularization Of LEft Main With Resolute onyX) A Multicenter Prospective Registry of the Onyx Resolute Stent for the Treatment of Unprotected Left Main Coronary Artery Disease.
Brief Title: The Rolex Registry (Revascularization Of LEft Main With Resolute onyX)
Acronym: Rolex
Status: Suspended | Type: Observational
Why Stopped: Waiting for a protocol amendment to extend follow-up lenght
Sponsor: University of Padova (Other)
Responsible Party: Sponsor
Other Study IDs: ROLEX_2017
Record Dates: First submitted 2017-10-06; First posted 2017-10-20 (Actual); Last update posted 2023-01-31 (Actual); Status verified 2023-01

CONDITIONS: Coronary Artery Disease
MeSH Terms: conditions — Coronary Artery Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

INTERVENTIONS:
Device: Resolute Onyx — Percutaneous coronary revascularization of patients with unprotected left main coronary artery disease up to intermediate anatomical complexity (defined by a SYNTAX score <33), must be performed with the exclusive use of drug-eluting stents of the Resolute Onyx TM family

SUMMARY:
The primary objective of this study is to assess the safety and efficacy of the new-generation zotarolimus-eluting stent Resolute Onyx in the treatment of unprotected left main coronary artery disease (ULMCAD), both isolated or in association with two- or three-vessel coronary artery disease.

DETAILED DESCRIPTION:
The ROLEX study is a prospective, non-randomized, European, multi-center registry.

Four hundred and fifty patients with unprotected left main coronary artery disease (ULMCAD) will be enrolled at up to 40 European sites. The main objective of the study is to assess the safety and efficacy of the new-generation zotarolimus-eluting stent Resolute Onyx in the treatment of ULMCAD, both isolated or in association with two- or three-vessel coronary artery disease

ELIGIBILITY:
Inclusion Criteria:

* Subject > 18 years old
* ULMCAD with angiographic diameter stenosis >50% (if 50-70% evidence of FFR <0.80 or IVUS minimal lumen area <6.0 mm2 is recommended.
* Silent ischemia, stable angina, unstable angina or non-ST elevation myocardial infarction
* Ability to provide written informed consent and comply with follow-up for at least 2 years.

Exclusion Criteria:

1. Clinical exclusion criteria:

   * Prior PCI on the left main trunk or prior CABG.
   * Concomitant indication to cardiac surgery (severe heart valve disease etc.)
   * Cardiogenic Shock (Killip>2)
   * Severe renal insufficiency (GFR <30 ml/min)
   * Known impaired left ventricular function (left ventricular ejection fraction <30%)
   * Inability to tolerate or comply with dual antiplatelet therapy for at least 1 year
   * Pregnancy or intention to become pregnant
   * Life expectancy less than 1 year
   * Other investigational drug or device studies that have not reached their primary endpoint
2. Angiographic exclusion criteria:

   * Left main diameter stenosis <50%
   * SYNTAX score >33

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Consecutive patients with unprotected left main coronary artery disease up to intermediate anatomical complexity (defined by a SYNTAX score <33), considered amenable for percutaneous coronary intervention (PCI).
Sampling Method: Non-Probability Sample
Enrollment: 450 (Actual)
Dates: Start 2017-11-01 (Actual); Primary Completion 2021-12-31 (Actual); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
target lesion failure | 12 months
  composite of cardiac death, target vessel myocardial infarction and ischemia-driven target lesion revascularization

CONTACTS AND LOCATIONS:
Overall Officials: Giuseppe Tarantini, MD, PhD, Principal Investigator — University of Padova
Locations (33):
- Italy (32):
  - Azienda Ospedale Università Padova, Padua, PD
  - ASP 1 Agrigento - Ospedale San Giovanni di Dio, Agrigento
  - Policlinico San Donato, Arezzo
  - Azienda Ospedaliera S.Anna e S.Sebastiano, Caserta
  - Ospedale Ferrarotto, Catania
  - Ospedale civile dell'Annunziata, Cosenza
  - Azienda Socio-Sanitaria Territoriale di Cremona, Cremona
  - Ospedale Santa Croce e Carle, Cuneo
  - Azienda Ospedaliera Grosseto, Grosseto
  - Ospedale Fazzi, Lecce
  - Ospedale Mater Salutis, Legnago
  - Azienda Ospedaliera Universitaria Policlinico G.Martino, Messina
  - Ospedale dell'angelo, Mestre
  - Centro cardiologico Monzino, Milan
  - Ospedale San Raffaele, Milan
  - Ospedale di Mirano, Mirano
  - Ospedali Riuniti Padova Sud "Madre Teresa di Calcutta", Monselice
  - Azienda Ospedaliera Universitaria Federico II, Napoli
  - Azienda Ospedliera Universitaria San Luigi Gonzaga, Orbassano
  - Policlinico San Marco, Osio Sotto
  - ARNAS Civico, Palermo
  - Fondazione IRCCS Policlinico San Matteo, Pavia
  - Ospedale Santo Spirito Santo, Pescara
  - Casa di Cura Dott. Pederzoli, Peschiera del Garda
  - Azienda Ospedaliera Bianchi Melacrino Morelli, Reggio Calabria
  - Ospedale degli infermi, Rivoli
  - Azienda Ospedaliera San Camillo Forlanini, Roma
  - Ospedale Sandro Pertini, Roma
  - Policlinico Gemelli, Roma
  - Azienda Ospedaliera Universitaria Senese, Siena
  - Ospedale Mauriziano Umberto I, Torino
  - Azienda Ospedaliera Universitaria Integrata Verona, Verona
- Hospital de Santa Cruz, Carnaxide, Portugal

REFERENCES:
- [Derived] Tarantini G, Fovino LN, Varbella F, Trabattoni D, Caramanno G, Trani C, De Cesare N, Esposito G, Montorfano M, Musto C, Picchi A, Sheiban I, Gasparetto V, Ribichini FL, Cardaioli F, Sacca S, Cerrato E, Napodano M, Martinato M, Azzolina D, Ando G, Mugnolo A, Caruso M, Rossini R, Passamonti E, Teles RC, Rigattieri S, Gregori D, Tamburino C, Burzotta F. A large, prospective, multicentre study of left main PCI using a latest-generation zotarolimus-eluting stent: the ROLEX study. EuroIntervention. 2023 Feb 6;18(13):e1108-e1119. doi: 10.4244/EIJ-D-22-00454. PMID 36043326